CLINICAL TRIAL: NCT01669200
Title: Effect of Medium Chain Triglyceride Oil Supplementation in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 12024
Record Dates: First submitted 2012-08-14; First posted 2012-08-20 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2013-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Oil (Placebo Comparator): Differential changes will be compared in the test group versus the control group at one month and six months with respect to BHB and insulin levels, and at six months with respect to cognitive scores.
  Interventions: Other: Placebo Oil
- Medium Chain Triglyceride Oil (Experimental): Differential changes will be compared in the test group versus the control group at one month and six months with respect to BHB and insulin levels, and at six months with respect to cognitive scores.
  Interventions: Other: Medium Chain Triglyceride Oil

INTERVENTIONS:
Other: Medium Chain Triglyceride Oil — Differential changes will be compared in the test group at one month and six months with respect to serum Beta-Hydroxybutyrate and insulin levels, and at six months with respect to cognitive scores.
  Arms: Medium Chain Triglyceride Oil
Other: Placebo Oil — Differential changes will be compared in the control group at one month and six months with respect to serum Beta-Hydroxybutyrate and insulin levels, and at six months with respect to cognitive scores.
  Arms: Placebo Oil

SUMMARY:
The primary aim of this study is to assess whether daily dosing with medium chain triglycerides in subjects with mild cognitive impairment (MCI) will improve cognitive performance.

DETAILED DESCRIPTION:
Twenty eligible subjects will be enrolled in the study that will consist of a baseline visit followed by six post-baseline visits. The control and placebo groups will each be comprised of ten subjects randomly assigned to the groups. The assessments at baseline will include concomitant medications, vital signs, height, and weight. In addition, subjects will complete a medical history questionnaire, and receive group instruction on incorporation of the study products into the diet from a registered dietitian. Study products will be dispensed at each visit in excess of requirements, and re-issued at every visit after measurement of the remaining product that subjects will be instructed to bring to every visit. The post-baseline study visits will include body weight and vital sign measurements, concomitant medications, dispensation of study products, group instruction by a registered dietitian, and an assessment for adverse events.

Between study visits the subjects will receive a telephone call from the study coordinator to encourage compliance with the diet, and to ask about any adverse events. The study visits will conclude at week 24. The psychological tests conducted by clinicians at screening will be repeated during the cognitive testing visit.

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female with a diagnosis of Mild Cognitive Impairment
2. Are 50 years of age or older

Exclusion Criteria:

1. Been on medication for Mild Cognitive Impairment less than 90 days
2. Major depression
3. Uncontrolled hypothyroidism
4. Known B12 deficiency
5. Hepatic (liver) disease or insufficiency

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Improvement in cognitive performance | Assess in subjects at Baseline to week 24 using different Cognitive testing scores.
  Daily dosing of in subjects with Medium Chain Triglyceride Oil will change cognition scores measured at baseline to the end of week 24 using cognitive testing results. (ADAS-Cog, Trails Making Test, Mini Mental State Exam, Digit Symbol Test and Short-Form 36 Health Survey).

SECONDARY OUTCOMES:
Serum Ketones | Baselines to 6 months
  A blood test will compare results looking for an increase of Beta-Hydroxybutyrate in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States